CLINICAL TRIAL: NCT02121678
Title: Effect of Resistance and Aerobic Exercise on Muscle Strength, Aerobic Capacity and Quality of Life in Patients Treated With Immunoglobulin for Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) or Multifocal Motor Neuropathy (MMN)
Brief Title: Effect of Resistance and Aerobic Exercise in CIDP or MMN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2013-200
Record Dates: First submitted 2014-02-17; First posted 2014-04-23 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; Multifocal Motor Neuropathy
Keywords: Resistance training; Aerobic exercise; Isokinetic muscle strength; Bicycle ergometry test; Subcutaneous immunoglobulin
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Run-in - Aerobic - Resistance (Experimental): * Week -12 to 0: Run-in period with no training
  * Week 0 to 12: Aerobic training on ergometer bicycle
  * Week 12 to 24: Resistance training with dumbbells
  Interventions: Other: Resistance training; Other: Aerobic training
- Run-in - Resistance - Aerobic (Experimental): * Week -12 to 0: Run-in period with no training
  * Week 0 to 12: Resistance training with dumbbells
  * Week 12 to 24: Aerobic training on ergometer bicycle
  Interventions: Other: Resistance training; Other: Aerobic training

INTERVENTIONS:
Other: Resistance training — Participants do resistance training of selected muscle groups. Resistance are predefined from 1-repetition max (1-RM) and increased during the 12 weeks of training:
  * Week 0-4: 70-80 % of 1-RM
  * Week 5-8: 75-86 % of 1-RM
  * Week 9-12: 80-92% of 1-RM
  Participants trains unilateral, the opposite site serves as reference.
  * MMN patients train elbow (flexion/extension) and wrist (flexion/extension)
  * CIDP patients train knee (flexion/extension) and elbow (flexion/extension)
Other: Aerobic training — Participants train on ergometer bicycle 2 times weekly increasing during the first weeks to 3 times weekly. Workload is measured before initiation and VO2-max, heart rate and blood pressure will be measured as well.
  Patients train with 60-75 % of VO2-max for 30 minutes per training session. They use heart rate monitor to store data.

SUMMARY:
Resistance and aerobic exercise has been shown to be effective for maintenance of muscle strength in patients with neuromuscular diseases.

Exercise in CIDP and MMN is sparsely described. The aim of the study is to evaluate changes in muscle strength during high intensive resistance training and changes in maximal oxygen consumption (VO2-max) during high intensive aerobic training in patients with CIDP or MMN in maintenance therapy with subcutaneous immunoglobulin.

The hypotheses are that muscle strength and VO2-max are significantly increased during the training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 80 years
* Diagnosed with definite or probable CIDP or definite or probable MMN fulfilling the European Federation of Neurological Sciences/Peripheral Nerve Society (EFNS/PNS) criteria
* Stable maintenance therapy with immunoglobulin (no change of dosage < 3 months before inclusion)
* Duration of CIDP or MMN > 6 months
* Negative result on a pregnancy test (HCG-based assay in urine) for women of childbearing potential and use of a reliable method of contraception for the duration of the study

Exclusion Criteria:

* Other cause of neuropathy (incl. pressure neuropathy)
* Exercise before enrolment (> 1 hour of exercise per week or > 4 km bicycling per day)
* Walking distance < 10 meter with or without aid
* Diabetes mellitus, severe cardiac or pulmonary disease, malignancies
* Known history of adverse reactions to Immunoglobulin A in other products
* Ongoing history of hypersensitivity or persistent reactions to blood or plasma derived products.
* History of malignancies of lymphoid cells and immunodeficiency with lymphoma
* Known liver function impairment (ALAT 3 times above upper limit of normal)
* Known protein-losing enteropathies or proteinuria.
* Known of renal function impairment (creatinine >120 micromol/L or creatinine >1.35 mg/dL), or predisposition for acute renal failure (e.g., any degree of pre-existing renal insufficiency or routine treatment with known nephritic drugs).
* Treatment with any investigational medicinal product within 3 months prior to first infusion of Gammanorm
* Known or suspected HIV, Hepatitis Virus C or B infection
* Pregnant or nursing women
* Planned pregnancy during course of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in isokinetic muscle strength | -12, 0, 6, 12 weeks or -12, 0, 12, 18, 24 weeks
  Changes in isokinetic muscle strength during resistance exercise. Four muscle groups bilateral are selected.
  CIDP: Knee flexion/extension Elbow flexion/extension MMN: Elbow flexion/extension Wrist flexion/extension
Changes in maximal oxygen consumption (VO2-max) | -12, 0, 6, 12 weeks or -12, 0, 12, 18, 24 weeks
  VO2-max are measured during the 12 weeks aerobic exercise session and at enrolment 12 weeks before start of exercise.
  VO2-max are measured while the participant running on a ergometer bicycle by accumulation of exhaled air

SECONDARY OUTCOMES:
Change in Medical Research Council (MRC) | -12, 0, 6, 12, 18, 24 weeks
Change in Overall Disability Sum Score (ODSS) | -12, 0, 6, 12, 18, 24 weeks
Change in 6-Minute Walk test | -12, 0, 6, 12 weeks or -12, 0, 12, 18, 24 weeks
Change in Quality of Life measured by The Short Form (36) Health Survey (SF-36) questionnaire | -12, 0, 6, 12, 18, 24 weeks
Change in Fatigue Severity Score (FSS) | -12, 0, 6, 12, 18, 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Neurology, Aarhus University Hospital, Aarhus C
  - Department of Neurology, Rigshospitalet, Copenhagen University Hospital, Copenhagen